CLINICAL TRIAL: NCT03638037
Title: Correlation Between Maternal Vitamin D Level And Preterm Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Dr- dina yahia mansour, Lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Other Study IDs: VD0074
Record Dates: First submitted 2018-08-13; First posted 2018-08-20 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Preterm Birth; Preterm Labor; Vitamin D Deficiency
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: 69 women, delivered preterm babies (less than 37weeks).
  Interventions: Diagnostic Test: Vitamin D measurement
- Control: 69 women, delivered at term (38-42 weeks) of full tem babies.
  Interventions: Diagnostic Test: Vitamin D measurement

INTERVENTIONS:
Diagnostic Test: Vitamin D measurement — Maternal serum 25- hydroxyl vitamin D level

SUMMARY:
Assessment of correlation between vitamin D level and prevalence of preterm births remains limited. The exact role of vitamin D in preterm birth has not yet been clearly defined ,where some studies showed vitamin D deficiency increased the risk of preterm birth while other studies found no correlation. In this study will try to continue research on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation.
* Maternal age: 20-35 years.

Exclusion Criteria:

1. Multi fetal pregnancy.
2. Anatomical or genetic defect of the fetus.
3. Iatrogenic preterm delivery.
4. Maternal medical disorder e.g diabetes millets (D.M).
5. Antepartum hemorrhage.
6. Hypertensive disorders.
7. Polyhydromins or oligolydromins
8. Premature rupture of membranes ± Chorioamnionitis
9. Incompetent cervix.
10. Post IVF.
11. Uterine Fibroid or malformation.

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women with singelton pregnancy
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2018-09-02 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with severe vitamin D deficiency | 3 months
  vitamin D deficiency defined as vitamin D level <10ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Maternity Hospital, Cairo, Egypt